CLINICAL TRIAL: NCT01007903
Title: Tai Chi Exercise in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Mind-Body Exercise for COPD: A Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Gloria Y. Yeh, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007P000065
Record Dates: First submitted 2009-11-03; First posted 2009-11-05 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Aquatic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Usual Care (No Intervention)
- Tai Chi (Experimental)
  Interventions: Behavioral: Tai Chi exercise

INTERVENTIONS:
Behavioral: Tai Chi exercise — 12-week tai chi exercise class
  Arms: Tai Chi

SUMMARY:
This is a pilot randomized controlled trial of feasibility and preliminary effects of a 12 week tai chi intervention vs. usual care in patients with chronic obstructive pulmonary disease

ELIGIBILITY:
Inclusion Criteria:

* physician diagnosis of COPD
* FEV1<65% of predicted and FEV1/FVC<0.70
* ≥45 years old

Exclusion Criteria:

* COPD exacerbation requiring ER visit or hospitalization within past month
* planned major pulmonary intervention in coming 3 months
* severe peripheral vascular disease/claudication or other physical condition precluding walk test
* inability to perform bicycle ergometry
* severe cognitive dysfunction (MMSE ≤ 24)
* inability to speak English
* current participation in a pulmonary rehabilitation or regular practice of tai chi

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10

PRIMARY OUTCOMES:
Study feasibility

SECONDARY OUTCOMES:
Quality of life
Exercise capacity

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Yeh, MD, MPH, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Yeh GY, Roberts DH, Wayne PM, Davis RB, Quilty MT, Phillips RS. Tai chi exercise for patients with chronic obstructive pulmonary disease: a pilot study. Respir Care. 2010 Nov;55(11):1475-82. PMID 20979675